CLINICAL TRIAL: NCT06464900
Title: Effects of a Health Education Intervention Based on the Behaviour Change Wheel on Fear of Hypoglycemia in Patients With Type 2 Diabetes Mellitus: a Randomized Controlled Study
Brief Title: Effects of a Health Intervention on Fear of Hypoglycemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhao Yueqi, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YZUHL20230040
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Health-Related Behavior; Health Education; Fear of Hypoglycemia; Impaired Awareness of Hypoglycemia; Self-Management; Type2 Diabetes Mellitus
Keywords: Behaviour Change Wheel; Health educational intervention; Fear of hypoglycaemic; Impaired awareness of hypoglycaemia; Medical support; Self-management attitude; Type 2 diabetes mellitus
MeSH Terms: conditions — Health Behavior; Health Education; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Care (Placebo Comparator): Implementation of routine diabetes health education.
  Interventions: Behavioral: Routine Care
- Based on BCW Theory of Health Education (Experimental): A FoH intervention program based on BCW theory was implemented on top of the routine care.
  Interventions: Behavioral: Based on BCW Theory of Health Education

INTERVENTIONS:
Behavioral: Routine Care — Provide patients with regular medication guidance, dietary guidance, exercise guidance and knowledge about diabetes mellitus and hypoglycaemia; test and record blood glucose regularly every day; answer patients' clinical questions and provide psychological support in a timely manner.
  Arms: Routine Care
Behavioral: Based on BCW Theory of Health Education — BCW theory was applied to analyse behaviour and develop interventions in terms of capability, motivation and opportunity. Capability: Intensive daily management of diabetes through intervention functions (education, training, persuasion, modelling) to change attitudes and habits, understand the negative consequences of fear of hypoglycaemia, improve hypoglycaemia awareness and self-regulation skills. Opportunity: Through the intervention function (education, training, realization) to improve the awareness of hypoglycemia awareness, timely detection of hypoglycemia. In the event of a hypoglycaemic event patients know how to deal with it. Motivation: Through intervention functions (environmental reconstruction, realisation) that take full account of external factors and their own opportunities. Glucose management through microsoft platforms, on-site teaching and coaching by specialist nurses to create opportunities for patients who can change excessive/avoidant behaviours.
  Arms: Based on BCW Theory of Health Education

SUMMARY:
To examine the effects of a health Education Intervention based on the Behaviour Change Wheel (BCW) theory on fear of hypoglycemia and relevant outcomes of type 2 diabetic patients.

DETAILED DESCRIPTION:
In this study, eligible participants were randomized in a 1:1 ratio into an intervention group (health education based on BCW theory given on top of regular diabetes health education) and a control group (regular diabetes health education), with a 4-week intervention period and a 8-week follow-up period, for a total of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Comply with the 2020 Chinese guidelines for the prevention and treatment of type 2 diabetes mellitus;
* Age ≥18 years;
* Duration of diabetes mellitus ≥1 year;
* FoH according to the elevated item endorsement criterion (E I criterion): ≥3 points on any item of the Hypoglycemic Fear-Worry Scale (HFS-WS);
* Patients who have the ability to listen, read, write, walk, and cooperate to complete the study;
* Patients who have a smart phone, and can skillfully use WeChat or telephone to communicate;
* Voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

* Patients with comorbid acute complications or other serious diseases or disorders of consciousness, such as diabetic hypertonic state, tumors, coma, etc;
* Patients with comorbid psychiatric diseases or taking psychotropic drugs;
* Patients who have recently or are participating in other studies on similar topics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Hypoglycemia fear survey | Baseline, 4 and 12 weeks post-intervention
  Fear of hypoglycemia (FoH) was assessed using the Hypoglycemic Fear Survey Scale (HFS), which consists of two subscales, the Hypoglycemic Fear Survey- Behavioral Scale (HFS-BS) and the Hypoglycemic Fear Survey-Worry Scale (HFS-WS). (1) The HFS-BS scale has 19 entries, using a 5-point Likert scale, with scores ranging from 1 ~ 5 in descending order, and a total score of 15 ~ 95, with higher scores indicating more obvious hypoglycemic fearful behaviors in patients. (2) HFS-WS has 13 entries, which were scored using a 5-point Likert scale, with scores ranging from 0 to 4 from low to high, and a total score of 0 ~ 52. The higher the score, the higher the degree of fear of hypoglycemia in patients. The two subscale scores were added together, and the higher the total score, the more severe the fear of hypoglycemia.

SECONDARY OUTCOMES:
Gold Rating | Baseline, 4 and 12 weeks post-intervention
  The Gold Score, first proposed by Professor Gold of the United Kingdom in 1994, is currently the most commonly used method of assessing Impaired Awareness of Hypoglycemia (IAH), which reflects the patient's awareness of hypoglycemia side by side. The method consists of a single question, "Do you know when your hypoglycemia began?" Answers are given on a 7-point Likert scale ranging from "1" (always aware) to "7" (never aware), with a score of 1-3 being considered normal self-awareness of hypoglycemia, and a score of ≥4 indicating the presence of IAH.
The Patients Assessment Chronic Illness Care( PACIC) | Baseline, 4 and 12 weeks post-intervention
  Used to assess the quality of care provided by healthcare organizations in the U.S. chronic disease management model. The scale is completed by patients to report the extent to which they have received care in the past 6 months consistent with the chronic disease management model and can be used to reflect the level of medical support provided to patients by chronic disease management organizations such as hospitals.The PACIC scale is divided into 5 dimensions and 20 questions, each of which is based on the use of a 5-dimensional model of care. 7~11), problem solving/coherence (entries 12~15), and follow-up/collaboration (entries 16~20), and each entry is rated on a 5-point Likert scale, with scores ranging from 1~5 from the lowest to the highest, and with scores closer to 5, the higher the evaluation of chronic disease management, and the more support the patient receives from healthcare professionals.
The self-management attitude scale for diabetes patients | Baseline, 4 and 12 weeks post-intervention
  The subscale has 5 entries to evaluate patients' attitudes toward diabetes health education, diet control, exercise, medication compliance, and blood glucose monitoring. A Likert 5-point scale was used, assigning values of 1.0, 0.8, 0.6, 0.4, 0.2 in descending order, and the total mean scores of the 5 entries (range 0.2-1.0) represented the self-management attitude scores. A total mean score of <3.0 indicates a poor self-management attitude, 3.0 to 4.25 indicates a moderate self-management attitude, and >4.25 indicates a good self-management attitude.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Yueqi, Master, Principal Investigator — Yangzhou University
Locations (1):
- Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No